CLINICAL TRIAL: NCT04537234
Title: Immunogenicity and Safety of a High-Dose Quadrivalent Influenza Vaccine in Subjects 65 Years of Age and Older in Taiwan
Brief Title: Study to Assess the Immune Response and the Safety Profile of a High-Dose Quadrivalent Influenza Vaccine (QIV-HD) Compared to a Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD) in Taiwanese Adults 65 Years of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QHD00023; U1111-1238-1970 (Other: UTN)
Record Dates: First submitted 2020-08-26; First posted 2020-09-03 (Actual); Results first posted 2021-11-08 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Influenza (Healthy Volunteers)
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was modified double-blind. The designated vaccine prepare(s)/administrator(s) would be unblinded given that the QIV-HD and QIV-SD vaccines had different dose volumes. Neither the participant nor the investigator nor the study staff in charge of vaccination was aware of which vaccine was administered (the syringes was masked to maintained the blinding of the participants and other members of the clinical site). The unblinded designated vaccine preparer(s)/administrator(s) was not involved in any of the blinded study assessments (eg, immunogenicity, safety).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) (Experimental): Participants received a single injection of 0.7 milliliters (mL) QIV-HD, intramuscularly (IM) at Day 0.
  Interventions: Biological: High-Dose Quadrivalent Influenza Vaccine
- Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD) (Active Comparator): Participants received a single injection of 0.5 mL QIV-SD, IM at Day 0.
  Interventions: Biological: Standard-Dose Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: High-Dose Quadrivalent Influenza Vaccine — Pharmaceutical form: Suspension for injection in pre-filled syringe,
  Route of administration: IM
  Other Names: Fluzone® High Dose, Efluelda™
  Arms: Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD)
Biological: Standard-Dose Quadrivalent Influenza Vaccine — Pharmaceutical form: Suspension for injection in pre-filled syringe,
  Route of administration: IM
  Other Names: AdimFlu-S (QIS)
  Arms: Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)

SUMMARY:
Primary Objective:

Immunogenicity: To describe the immune response induced by high-dose quadrivalent influenza vaccine (QIV-HD) and AdimFlu-S (QIS) by hemagglutinin inhibition (HAI) measurement method in all participants.

Safety: To describe the safety profile of all participants in each study groups.

DETAILED DESCRIPTION:
The duration of each participant's participation was approximately 28 days (Day 0 through Day 28 [+ 7 days]).

ELIGIBILITY:
Inclusion criteria :

* 65 years and older on the day of inclusion.
* Able to attend all scheduled visits and complied with all study procedures.

Exclusion criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the study vaccination or planned receipt of any vaccine prior to Visit 2.
* Previous vaccination against influenza (in the preceding 6 months) with either the study vaccine or another vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the study or to a vaccine containing any of the same substances.
* Thrombocytopenia, bleeding disorder, or receipt of anticoagulants that based on Investigator's judgment contraindicate intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion.
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature greater than or equal to [>=] 38.0 degree Celsius). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Personal or family history of Guillain-Barré syndrome.
* Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that was stable at the time of vaccination in the absence of therapy and participants who had a history of neoplastic disease and had been disease free for >=5 years).
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse) of the Investigator or employee with direct involvement in the proposed study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 165 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- Taiwan (4):
  - Investigational Site Number 1580004, Taichung
  - Investigational Site Number 1580001, Taipei
  - Investigational Site Number 1580002, Taipei
  - Investigational Site Number 1580003, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Chen JY, Hsieh SM, Hwang SJ, Liu CS, Li X, Fournier M, Yeh TY, Yin JK, Samson SI. Immunogenicity and safety of high-dose quadrivalent influenza vaccine in older adults in Taiwan: A phase III, randomized, multi-center study. Vaccine. 2022 Oct 26;40(45):6450-6454. doi: 10.1016/j.vaccine.2022.09.078. Epub 2022 Oct 7. PMID 36216650
- See also: QHD00023 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25342&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 active centers in Taiwan. A total of 165 participants were enrolled and randomized between 10 November 2020 to 12 January 2021.
Pre-assignment Details: A total of 165 participants were vaccinated in the study.
Period: Overall Study
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
Started | 82 | 83
Completed | 80 | 83
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD): Participants received a single injection of 0.7 mL QIV-HD, IM at Day 0.
- Total: Total of all reporting groups
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD) | Total
Number analyzed (Participants) | 82 | 83 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (5.37) | 71.4 (5.71) | 71.4 (5.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 93
  Male | 35 | 37 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 82 | 83 | 165
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies at Day 0
Description: GMTs of anti-influenza antibodies were measured using hemagglutination inhibition (HAI) assay for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria Lineage), and B2 (B Yamagata Lineage). Titers were expressed in terms of 1/dilution.
Time Frame: Day 0 (pre-vaccination)
Population: Analysis was performed on the full analysis set (FAS) that included randomized participants who received one of the study vaccine and had a post-vaccination blood sample. Participants were analyzed according to the vaccine group to which they were randomized.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
Number analyzed (Participants) | 80 | 83
titers
  A/H1N1 | 23.6 [18.1 to 30.6] | 24.1 [18.5 to 31.5]
  A/H3N2 | 111 [78.4 to 156] | 169 [120 to 238]
  B1 | 88.0 [66.7 to 116] | 98.2 [76.6 to 126]
  B2 | 149 [111 to 199] | 160 [121 to 211]

2. Primary Outcome: Geometric Mean Titers of Influenza Vaccine Antibodies at Day 28
Description: GMTs of anti-influenza antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage). Titers were expressed in terms of 1/dilution.
Time Frame: Day 28 (post-vaccination)
Population: Analysis was performed on FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
Number analyzed (Participants) | 80 | 83
titers
  A/H1N1 | 283 [221 to 364] | 109 [78.2 to 151]
  A/H3N2 | 643 [522 to 791] | 427 [324 to 563]
  B1 | 812 [645 to 1023] | 324 [253 to 414]
  B2 | 707 [595 to 840] | 361 [290 to 450]

3. Primary Outcome: Geometric Mean Titers Ratio (GMTR) of Influenza Vaccine Antibodies
Description: GMTRs of anti-influenza antibodies were measured by using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage). GMTRs were calculated as the ratio of GMTs post-vaccination (on Day 28) and pre-vaccination (on Day 0).
Time Frame: Day 0 (pre-vaccination), Day 28 (post-vaccination)
Population: Analysis was performed on FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
Number analyzed (Participants) | 80 | 83
ratio
  A/H1N1 | 12.0 [9.09 to 15.9] | 4.50 [3.47 to 5.82]
  A/H3N2 | 5.81 [4.28 to 7.87] | 2.53 [1.87 to 3.41]
  B1 | 9.23 [7.00 to 12.2] | 3.30 [2.48 to 4.39]
  B2 | 4.76 [3.65 to 6.21] | 2.26 [1.76 to 2.89]

4. Primary Outcome: Percentage of Participants Achieving Seroconversion Against Influenza Virus Antigens
Description: Anti-influenza antibodies were measured by HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage). Seroconversion was defined as either a pre-vaccination HAI titer less than (<) 10 (1/dilution) at Day 0 and a post-vaccination titer greater than or equal to (>=) 40 (1/dilution) at Day 28 or a pre-vaccination titer >=10 (1/dilution) at Day 0 and a >= four-fold increase in post-vaccination titer at Day 28.
Time Frame: Day 28 (post-vaccination)
Population: Analysis was performed on FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
Number analyzed (Participants) | 80 | 83
percentage of participants
  A/H1N1 | 86.3 [76.7 to 92.9] | 50.6 [39.4 to 61.8]
  A/H3N2 | 61.3 [49.7 to 71.9] | 28.9 [19.5 to 39.9]
  B1 | 78.8 [68.2 to 87.1] | 37.3 [27.0 to 48.7]
  B2 | 50.0 [38.6 to 61.4] | 24.1 [15.4 to 34.7]

5. Primary Outcome: Percentage of Participants With Antibody Titers >=40 (1/Dilution) at Day 0
Description: Antibody titer was measured by using HAI assay method for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage).
Time Frame: Day 0 (pre-vaccination)
Population: Analysis was performed on FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
Number analyzed (Participants) | 80 | 83
percentage of participants
  A/H1N1 | 33.8 [23.6 to 45.2] | 36.1 [25.9 to 47.4]
  A/H3N2 | 76.3 [65.4 to 85.1] | 84.3 [74.7 to 91.4]
  B1 | 81.3 [71.0 to 89.1] | 85.5 [76.1 to 92.3]
  B2 | 85.0 [75.3 to 92.0] | 86.7 [77.5 to 93.2]

6. Primary Outcome: Percentage of Participants With Antibody Titers >=40 (1/Dilution) at Day 28
Description: Antibody titer was measured using HAI assay method for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage).
Time Frame: Day 28 (post-vaccination)
Population: Analysis was performed on FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
Number analyzed (Participants) | 80 | 83
percentage of participants
  A/H1N1 | 97.5 [91.3 to 99.7] | 79.5 [69.2 to 87.6]
  A/H3N2 | 100 [95.5 to 100] | 96.4 [89.8 to 99.2]
  B1 | 98.8 [93.2 to 100] | 98.8 [93.5 to 100]
  B2 | 100 [95.5 to 100] | 100 [95.7 to 100]

7. Primary Outcome: Number of Participants With Immediate Unsolicited Systemic Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a patient or in a clinical investigation participant administered a medicinal product and which did not had any causal relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination. All participants were observed for 30 minutes after vaccination, and any unsolicited systemic AEs occurred during that time were recorded as immediate unsolicited AEs in the CRB.
Time Frame: Within 30 minutes post-vaccination
Population: Analysis was performed on the safety analysis set (SafAS) that included participants who had received one of the study vaccines and had any safety data available; and were analyzed according to the vaccine they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
Number analyzed (Participants) | 82 | 83
Participants | 0 | 0

8. Primary Outcome: Number of Participants With Solicited Injection Site and Systemic Reactions
Description: A solicited reaction was an "expected" adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the protocol and CRB and considered as related to the product administered. Solicited injection site reactions included pain, erythema, swelling, induration, and bruising. Solicited systemic reactions included fever, headache, malaise, myalgia and shivering.
Time Frame: Within 7 days post-vaccination
Population: Analysis was performed on the SafAS. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
Number analyzed (Participants) | 82 | 83
Participants
  Injection site Pain | 37 | 30
  Injection site Erythema | 8 | 7
  Injection site Swelling | 8 | 2
  Injection site Induration | 8 | 2
  Injection site Bruising | 0 | 0
  Fever: number analyzed (Participants) | 80 | 83
  Fever | 1 | 0
  Headache | 9 | 4
  Malaise | 9 | 7
  Myalgia | 22 | 10
  Shivering | 3 | 3

9. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An AE was any untoward medical occurrence in a patient or in a clinical investigation participant administered a medicinal product and which did not had any causal relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRB in terms of diagnosis and/or onset window post-vaccination.
Time Frame: Within 28 days post-vaccination
Population: Analysis was performed on the SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
Number analyzed (Participants) | 82 | 83
Participants | 8 | 12

10. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Including Adverse Event of Special Interest (AESIs)
Description: An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. AESIs was defined as event for which ongoing monitoring and rapid communication by the investigator to the sponsor was done.
Time Frame: From Day 0 up to 28 days post-vaccination
Population: Analysis was performed on the SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
Number analyzed (Participants) | 82 | 83
Participants
  SAE | 0 | 0
  AESIs | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AEs were collected from Day 0 (post-vaccination) up to 28 days post-vaccination. Solicited reaction data were collected up to Day 7 post-vaccination. SAE data were collected from Day 0 (post-vaccination) up to 28 days post-vaccination.
Description: A solicited reaction was an "expected" adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the protocol and CRB and considered as related to the product administered. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the CRB in terms of diagnosis and/or onset window post-vaccination. Analysis was performed on SafAS.
Arm/Group | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD)
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/83
Other Adverse Events (participants affected / at risk) | 46/82 | 35/83
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) (N=82) | Group 2: Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD) (N=83)
Injection Site Erythema (General disorders) | 8 (8) | 7 (7)
Injection Site Induration (General disorders) | 8 (8) | 2 (2)
Injection Site Pain (General disorders) | 37 (37) | 30 (30)
Injection Site Swelling (General disorders) | 8 (8) | 2 (2)
Malaise (General disorders) | 9 (9) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 22 (22) | 10 (10)
Headache (Nervous system disorders) | 9 (9) | 5 (5) — Headache events that occurred after 7 days post-vaccination were considered as unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT04537234/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT04537234/SAP_001.pdf